CLINICAL TRIAL: NCT04027114
Title: Individualized Physiotherapy and Activity Coaching for Multiple Sclerosis (IPAC-MS): A Randomised Controlled Trial
Brief Title: Individualized Physiotherapy and Activity Coaching for Multiple Sclerosis
Acronym: IPAC-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (SHRF) (Unknown); Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Principal Investigator, Sarah Donkers, Assistant Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Bio-1019
Record Dates: First submitted 2019-07-10; First posted 2019-07-19 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Multiple Sclerosis
Keywords: randomized controlled trial; multiple sclerosis; physiotherapy; behaviour change; physical activity; exercise; disability progression; walking function
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioural Physical Activity (PA) intervention (Experimental)
  Interventions: Behavioral: Individualized behavioural physical activity intervention
- Wait list control (No Intervention)

INTERVENTIONS:
Behavioral: Individualized behavioural physical activity intervention — • The intervention involves a tailored physiotherapy (PT) intake that will serve as the foundation for the individualized approach. Participants' individual attributes and physical activity needs, including a general PT assessment will occur initially. Over the next 12 months, participants will receive individualized PT coaching and a physical activity plan plus access to educational literature that outlines methods and benefits of exercise. An estimated 15 hours of PT contact hours per participant is anticipated and the specifics of each encounter will be documented.
  Arms: Behavioural Physical Activity (PA) intervention

SUMMARY:
Multiple Sclerosis (MS) is a chronic neurological disease that places a high burden on patients, families and society. Physical activity in MS is associated with improved fitness, symptoms, and function, fewer relapses, and fewer brain lesions on MRI. Saskatchewan has one of the highest rates of MS worldwide, and a recent survey estimated approximately 80% of persons living with MS are not sufficiently active for health benefits. Individuals living with MS recognize the importance of physical activity, but often indicate a lack support, including limited access to professionals knowledgeable about both MS and physical activity. There is a need to identify effective interventions for improving activity levels safely and appropriately. Behaviour change strategies target specific behaviours involved in increasing and maintaining physical activity. The primary objective of this project is to determine if individualized behaviour change strategies delivered by neurophysiotherapists increases physical activity in MS. Participants will be randomly assigned into two groups. The intervention group will receive individualized behaviour change strategies delivered through the support of neurophysiotherapists for 12 months. The wait-list control group will receive usual care for 12 months, and then be offered the intervention for a 6-month period at the end of the study period. The long-term goal of this research is to help decrease the burden of MS by identifying new opportunities for increasing physical activity.

ELIGIBILITY:
Inclusion Criteria:

* clinically definite MS (diagnosed by a neurologist)
* patient determined disease steps (PDDS) less than or equal to 6 (i.e. not wheel-chair bound)
* GLTEQ<24 (not active enough for health benefits)

Exclusion Criteria:

* medical instability (PAR-Q moderate-high risk of exercise-related harm)
* persons unable to provide consent
* persons under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Godin Leisure Time Exercise Questionnaire (GLTEQ) Score | baseline to 12 months
  change in physical activity level. The GLTEQ is a 4-item self-administered questionnaire with the first three questions seeking information on the number of times one engages in mild, moderate and strenuous activity in bouts of at least 15 min duration in a typical week. Total leisure activity score is then calculated based on number of bouts at each intensity multiplied by 3, 5, and 9 metabolic equivalents and summed. A higher score means more physically active.

SECONDARY OUTCOMES:
Multiple Sclerosis Impact Scale version 2 (MSIS-29 v2) | baseline to 12 months
  change in patient-reported disease-related symptoms measured using MSIS-29 v2 scale. MSIS-29 assess the impact of MS on health related quality of life in terms of physical and psychological well-being. The MSIS-29 v2 is a 29 item self-administered questionnaire. 20 items are associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 4 response options: 1 "not at all" to 4"extremely". Min score=29, max =116 with a higher value indicating more severely impacted
Multiple Sclerosis Self Efficacy Scale (MSSE) | baseline to 12 months
  change in patient-reported level of confidence regarding components of disease management. The MSSE has 18 items represented by two subscales of Function (9 items) and Control (9 items). Participants rate their confidence from 10-100 where 10 has an anchor of very uncertain, 50 moderately certain, and 100 very certain. A higher score meaning more confident/higher self-efficacy.
Interviews and Exit surveys | after intervention (at 12 month point for intervention group and 18 month for wait-list control) group
  experience of participants and interventionists
Intervention Description | after intervention (at 12 month point for intervention group and 18 month for wait-list control group)
  a description of interventionist contact time with participant and frequency, method and types of services provided

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Donkers SJ, Evans C, Levin MC, Ives K, Le H, Lim HJ, Knox KB. Individualized Physiotherapy and Activity Coaching in Multiple Sclerosis (IPAC-MS): Results of a Randomized Controlled Trial. Arch Phys Med Rehabil. 2025 Aug;106(8):1145-1154. doi: 10.1016/j.apmr.2025.02.005. Epub 2025 Feb 15. PMID 39961428
- [Derived] Goulding FL, Evans CD, Knox KB, Lim HJ, Levin MC, Donkers SJ. Individualised behaviour change strategies for physical activity in multiple sclerosis (IPAC-MS): protocol for a randomised controlled trial. Trials. 2019 Dec 2;20(1):664. doi: 10.1186/s13063-019-3768-7. PMID 31791380